CLINICAL TRIAL: NCT03098186
Title: TXT2HEART COLOMBIA: Evaluation of the Efficacy and Safety of Text Messages to Improve Adherence to Cardiovascular Medications in Secondary Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University College, London (Other); Universidad Pontificia Bolivariana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 416
Record Dates: First submitted 2017-03-10; First posted 2017-03-31 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Cardiovascular Disease
Keywords: Medication adherence; mHealth
MeSH Terms: conditions — Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: TX2THeart-Colombia is a single-blind trial. The laboratory personnel in charge of measurement LDL-C and 11 dhTxB2 levels will not have access to treatment allocation and they will only have access to internal numerical ID variable. The laboratory results will be conducted once trial follow-up is completed, and results will be sent directly to the database manager, who will link the results to the existing database. The staff in charge of measurement blood-pressure and heart rate will not have access to information on treatment allocation. Measurement of blood pressure and heart rate will be the first activity to be conducted with participants in visits 1 and 3 to minimize any potential subconscious bias introduced as a consequence of patients inadvertently revealing to trial staff the treatment allocation. The only person who will have access to the information of the participants is the engineer in charge of the management of Dimagi-Commcare Plataform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention SMS (Active Comparator): 1. SMS aimed to improved adherence to medications used in secondary prevention of cardiovascular disease.
  2. Control SMS: SMS to thanks for participation in the trial and reminders of trial appointments.
  Interventions: Behavioral: Intervention SMS
- Control SMS (Placebo Comparator): SMS to thanks for participation in the trial and reminders of trial appointments.
  Interventions: Behavioral: Control SMS

INTERVENTIONS:
Behavioral: Intervention SMS — The active treatment will consist of SMS that are aimed to modified behavioral factors associated with poor adherence to cardiovascular medications used in secondary prevention. The SMS will be delivered daily during the first month, increasing one day of interval for each week during the second month , and weekly thereafter until end of month 12th. In addition, they will receive SMS thanking for their participation in the trial, reminders of trial appointment and informing if they have changed contact details. The frequency of this SMS will be monthly.
  Arms: Intervention SMS
Behavioral: Control SMS — Participants will only receive the SMS thanking for their participation in the trial, reminders of trial appointment and informing if they have changed contact details. The frequency of this SMS will be monthly.
  Arms: Control SMS

SUMMARY:
Purpose of the trial: To evaluate the efficacy and safety of an intervention with SMS messages delivered by mobiles phones to improve adherence to cardiovascular medications in patients with atherosclerotic cardiovascular disease (ASCVD).

Trial design: Two-parallel arm, single-blind, individually randomized controlled trial.

Primary endpoint: Differences in changes (baseline minus 12 months) of: Low density lipoprotein cholesterol (LDL-C), Systolic Blood pressure and Heart Rate.

Secondary endpoints: Differences in the changes (baseline minus 12-months) of: (i) adherence to cardiovascular medications used in secondary prevention measured by MARS-5 questionnaire; and (ii) Urinary levels of 11 dh-TxB2, Rates of composite end-point of cardiovascular death and hospitalization due to cardiovascular disease up to 12 months, Rates of composite of non-cardiovascular death or hospitalizations due to non-cardiovascular disease up to 12 months and Adverse events: traffic accidents and injuries while reading SMS related to the trial.

Duration of follow-up: 12 months

Trial treatment:

Intervention: The active treatment will consist of SMS that are aimed to modified behavioral factors associated with poor adherence to cardiovascular medications used in secondary prevention. The SMS will be delivered daily during the first month, increasing one day of interval for each week during the second month, and weekly thereafter until end of month 12th. In addition, they will receive SMS thanking for their participation in the trial, reminders of trial appointment and informing if they have changed contact details. The frequency of this SMS will be monthly.

Control: participants will only receive the SMS thanking for their participation in the trial, reminders of trial appointment and informing if they have changed contact details. The frequency of this SMS will be monthly.

Expected sample size, enrollment and expected number of centers:

Sample size = 1600 Recruitment start date: March , 2017 Recruitment end date: September, 2017 Follow-up end date: March, 2018 Number of centers: 1

Statistical considerations:

* Intention to treat analysis
* The trial has >90% power (2 sided alpha= 0.05) to detect a reduction in LDL-C as low as 5.1 mg/dl, under the assumption that SMS will increase adherence to statins by 7%.
* The primary outcomes will be analyzed using ANCOVA.

Partially Financed by COLCIENCIAS Code: 656672553352

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* History of at least one of the following arterial occlusive events:

  * acute coronary syndrome (unstable angina, acute myocardial infarction with or without ST elevation),
  * stable angina,
  * ischemic cerebrovascular disease,
  * peripheral arterial disease or
  * coronary revascularization (coronary artery bypass surgery (CABG) or percutaneous transluminal coronary angioplasty (PTCA).
* Own at least one mobile phone
* Ability to read and understand text messages (SMS)
* Intention to stay in the country of recruitment during the next 12 months

Exclusion Criteria:

* Contraindication to take all cardiovascular medications used in secondary prevention.
* Participation in another randomized clinical trial that could interfere with adherence to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Differences in physiological variables depending on taking medications: low density lipoprotein cholesterol | Baseline and 12 months
  Low density lipoprotein cholesterol (LDL-C) mg/dl
Differences in physiological variables depending on taking medications: Systolic Blood pressure | Baseline and 12 months
  Systolic Blood pressure mmHg
Differences in physiological variables depending on taking medications: Heart Rate | Baseline and 12 months
  Heart Rate: Heartbeats per minute

SECONDARY OUTCOMES:
Changes in self-reported adherence and recurrence of new cardiovascular and adverse events. | Baseline and 12 months
  Adherence to cardiovascular medications used in secondary prevention measured by MARS-5 questionnaire
Urinary levels of 11 dh-TxB2 | Baseline and 12 months
  Changes in Urinary levels of 11 dh-TxB2 pg/dl
Death due to cardiovascular disease | Baseline and 12 months
  Rate of death due to cardiovascular disease.
Hospitalization due to cardiovascular disease | Baseline and 12 months
  Rate of hospitalization due to cardiovascular disease.
Death due to non-cardiovascular disease | Baseline and 12 months
  Rate of death due to non-cardiovascular disease.
Hospitalization due to non-cardiovascular disease | Baseline and 12 months
  Rate of hospitalizations due to non-cardiovascular disease.
Adverse events | Baseline and 12 months
  Traffic accidents and injuries while reading SMS related to the trial. (Percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Casas, PhD, Study Chair — University College, London; Pablo A Perel, PhD, Study Chair — London School of Hygiene and Tropical Medicine; Norma C Serrano, MsC, Study Director — Fundación Cardiovascular de Colombia; Anderson Bermon, MsC, Principal Investigator — Fundación Cardiovascular de Colombia; Ana F Uribe, PhD, Principal Investigator — Universidad Pontificia Bolivariana
Locations (1):
- Fundación Cardiovascular de Colombia, Floridablanca, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bermon A, Uribe AF, Perez-Rivero PF, Prieto-Merino D, Saaibi JF, Silva FA, Canon DI, Castillo-Gonzalez KM, Caceres-Rivera DI, Guio E, Meneses-Castillo KJ, Castillo-Meza A, Atkins L, Horne R, Murray E, Serrano NC, Free C, Casas JP, Perel P. Efficacy and Safety of Text Messages Targeting Adherence to Cardiovascular Medications in Secondary Prevention: TXT2HEART Colombia Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Jul 28;9(7):e25548. doi: 10.2196/25548. PMID 34319247
- [Derived] Bermon A, Uribe-Rodriguez AF, Perez-Rivero PF, Prieto-Merino D, Caceres Rivera DI, Guio E, Atkins L, Horne R, Murray E, Serrano Diaz NC, Free C, Perel P, Casas JP. Evaluation of the efficacy and safety of text messages targeting adherence to cardiovascular medications in secondary prevention: the txt2heart Colombia randomised controlled trial protocol. BMJ Open. 2019 Dec 8;9(12):e028017. doi: 10.1136/bmjopen-2018-028017. PMID 31818831